CLINICAL TRIAL: NCT01466751
Title: Neurobehavioral Intervention as a Novel Treatment Approach for Emotion-Regulatory Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Etkin, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-19338
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Anxiety; Depression
Keywords: Computerized neurobehavioral intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Engaging computerized tasks (Active Comparator): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention
- Neurobehavioral computerized tasks (Experimental): Participants will log into a personalized website and engage in computerized tasks online.
  Interventions: Behavioral: Computerized Neurobehavioral Intervention

INTERVENTIONS:
Behavioral: Computerized Neurobehavioral Intervention — Targeted, computerized interventions completed from the participants' own home on a computer.

SUMMARY:
The present study will explore the effectiveness of a computer based neurobehavioral intervention in alleviating symptoms and improving emotion regulation in psychiatric populations. It will increase understanding of psychopathology at a neural-circuit level and aid development of new non-pharmacological treatment for emotion regulatory deficits.

ELIGIBILITY:
Inclusion Criteria:

* current anxiety or depression symptoms
* internet access

Exclusion Criteria:

* lifetime psychotic disorder, past-year substance dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Fonzo, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neurobehavioral Computerized Tasks | Engaging Computerized Tasks
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engaging Computerized Tasks | Neurobehavioral Computerized Tasks | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10) | 36 (12) | 35.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 9 | 8 | 17
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time to Facial Affect Identification During Emotional Conflict
Description: A standardized set of facial emotions (fear and happy) were presented for a duration of about 1 second in quick succession (a new face every 3-5 seconds). Across each face was written an emotional word ("FEAR" or "HAPPY"), which could be either congruent or incongruent with the facial expression. The participant was instructed to identify the facial emotion as quickly as possible and ignore the overlaid emotion word. The outcome measure of interest was the average speed (across all trials presented) within which an individual could correctly identify the facial emotion as a function of time (pre or post-intervention), treatment arm (control or intervention), facial affect (fear or happy), and congruency of word and facial affect (congruent or incongruent).
Time Frame: Baseline, 3-month
Population: Participants who complete the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Engaging Computerized Tasks | Neurobehavioral Computerized Tasks
Number analyzed (Participants) | 12 | 12
milliseconds
  Baseline Congruent Fear | 802.15 (155.14) | 889.14 (135.65)
  Baseline Incongruent Fear | 848.79 (142.18) | 937.97 (151.94)
  Baseline Congruent Happy | 764.08 (130.52) | 868.45 (131.05)
  Baseline Incongruent Happy | 830.06 (142.29) | 961.49 (134.32)
  3 Month Congruent Fear | 814.58 (158.56) | 872.84 (178.04)
  3 Month Incongruent Fear | 863.80 (144.65) | 909.89 (193.45)
  3 Month Congruent Happy | 796.54 (130.62) | 824.36 (196.77)
  3 Month Incongruent Happy | 878.40 (175.54) | 890.90 (196.22)
Statistical Analysis 1: Comparison: Engaging Computerized Tasks vs Neurobehavioral Computerized Tasks; A linear mixed model was utilized to test the null hypothesis that the intervention groups would show equivalent performance change on the outcome measure from baseline to the 3 month time points; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — A-priori threshold for statistical significance: p < 0.05. No correction for multiple comparisons. The omnibus effect from the linear mixed model for the Treatment Arm x Time Interaction was utilized to establish significance of the effect; Numerator degrees of freedom=1, Denominator degrees of freedom = 168; Type III Tests of Fixed Effects = 8.687

2. Primary Outcome: Amygdala Blood Oxygenation-level Dependent Response (BOLD) Activation to Face Affect Identification During Emotional Conflict
Description: The degree of differential BOLD signal change (T2*-weighted contrast in a defined region of the brain as measured by functional magnetic resonance imaging) within each individual, averaged across trials, during facial affect identification (fear or happy) and induction of emotional conflict (when the emotion word "FEAR" or "HAPPY" was either congruent or incongruent with the facial expression). We examined the differential degree of amygdala BOLD signal change as a function of emotion type (fear or happy), congruency (congruent or incongruent), and hemisphere (left or right) at baseline and 3 months.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: Percentage of BOLD signal change
Arm/Group | Neurobehavioral Computerized Tasks | Engaging Computerized Tasks
Number analyzed (Participants) | 14 | 14
Percentage of BOLD signal change
  Baseline Left Amygdala Fear | 0.21 (0.93) | 0.16 (0.54)
  Baseline Left Amygdala Happy | 0.25 (1.05) | -0.29 (0.79)
  Baseline Right Amygdala Fear | 0.04 (1.24) | 0.02 (0.60)
  Baseline Right Amygdala Happy | -0.30 (0.86) | -0.23 (0.85)
  3 Month Left Amygdala Fear | 0.13 (0.85) | 0.38 (0.79)
  3 Month Left Amygdala Happy | -0.03 (0.76) | 0.18 (1.02)
  3 Month Right Amygdala Fear | 0.05 (0.66) | 0.21 (0.92)
  3 Month Right Amygdala Happy | -0.10 (0.85) | 0.05 (0.85)
Statistical Analysis 1: Comparison: Neurobehavioral Computerized Tasks vs Engaging Computerized Tasks; A linear mixed model was used to test the null hypothesis that the two treatment groups would display no differential changes in amygdala BOLD signal from baseline to 3 months as a main effect or in interaction with facial affect type (fear or happy) or by brain hemisphere (left or right); Test type: Superiority or Other; p = 0.156, Mixed Models Analysis — No adjustment for multiple comparisons. The a priori threshold was: p < 0.05; Numerator degrees of freedom: 1, Denominator degrees of freedom: 168; Type III Tests of Fixed Effects = 2.032

ADVERSE EVENTS:
Arm/Group | Engaging Computerized Tasks | Neurobehavioral Computerized Tasks
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No